CLINICAL TRIAL: NCT04948385
Title: Can Patients Who Have Undergone a Digestive Endoscopy Under Deep Sedation Drive Their Vehicle as Soon as a Post-Anesthetic Discharge Scoring System (PADDS) Equal to 9 is Obtained ?
Brief Title: Driving Performance After Deep Sedation for Outpatient Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Claude Hallet, Principal investigator, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B7007201938885
Record Dates: First submitted 2021-06-03; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Driving Impaired
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Active Comparator): Deep sedation for digestive endoscopy.
  Interventions: Drug: Propofol
- Escorts (Other): Accompanying persons are the adults who accompany the patients home. They do not receive any medication or intervention.
  Interventions: Procedure: No sedation

INTERVENTIONS:
Drug: Propofol — deep sedation with propofol +/- adjuvants such as midazolam, sufentanil, lidocaine and/or dehydrobenperidol
  Arms: Patients
Procedure: No sedation — No sedation
  Arms: Escorts

SUMMARY:
Many drugs used during anesthesia can reduce alertness and therefore present potential risks when driving a vehicle (risk of accident). Some scientific societies recommend not driving for 12 to 24 hours after sedation or general anesthesia. However, there are conflicting data in the literature showing that general anesthesia in healthy volunteers does not impair driving ability as early as 2 hours after the end of anesthesia.

This need not to drive requires the outpatient to have an escort. Unfortunately, some patients find it difficult to benefit from an adult escort, which can lead to last minute cancellations, absences or the need for a classic overnight hospital stay.

The main objective of the study is to compare with a simulator the driving performances of patients who have benefited from deep sedation for an outpatient endoscopic digestive procedure when they have met the discharge criteria to the performances of their escorts in order to determine if the conditions are as safe to let them drive home.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a driver license

Exclusion Criteria:

* Unavailabilty of the escort for the duration of the examination
* No driving for the past 5 years
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Travel time | until the end of the driving test, an average of 1 hour.
Number of collisions | until the end of the driving test, an average of 1 hour.
Number of collisions with a pedestrian | until the end of the driving test, an average of 1 hour.
Number of times over the speed limit | until the end of the driving test, an average of 1 hour.
Percentage of speeding time | until the end of the driving test, an average of 1 hour.
Percentage of speeding distance | until the end of the driving test, an average of 1 hour.
Number of speeding ticket | until the end of the driving test, an average of 1 hour.
Number of crossings of the median line | until the end of the driving test, an average of 1 hour.
Number of passages on the shoulder | until the end of the driving test, an average of 1 hour.
Percentage of time out of traffic lane | until the end of the driving test, an average of 1 hour.
Percentage of distance out of traffic lane | until the end of the driving test, an average of 1 hour.
Number of broken stops | until the end of the driving test, an average of 1 hour.
Number of stops at traffic lights | until the end of the driving test, an average of 1 hour.
Number of traffic light ticket | until the end of the driving test, an average of 1 hour.

SECONDARY OUTCOMES:
Karolinska Sleepiness Scale (KSS) | Within 30 minutes before driving test with simulator
  9-points scale : 1 (extremely alert) to 9 (very sleepy)
Karolinska Sleepiness Scale (KSS) | Within 10 minutes after driving test with simulator
  9-points scale : 1 (extremely alert) to 9 (very sleepy)
Beck II Depression inventory score (BDI-II) | Within 30 minutes before driving test with simulator
  21 items - 0 to 3 points by item - 0 (minimal) to 63 (severe depression)
STOP-Bang questionnaire (Snoring, Tired, Observed, Pressure, Body Mass index > 35, Age, Neck size, Gender) | Within 30 minutes before driving test with simulator
  0 to 8 points (0 = low risk to 8 = high risk of sleep apnea)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire de Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No